CLINICAL TRIAL: NCT00974948
Title: A Randomized, Double Blind, Sham-Controlled Trial of EUS-Guided Celiac Plexus Neurolysis (EUS-CPN) for Pain Due to Newly Diagnosed, Inoperable Pancreatic Cancer
Brief Title: Trial of Endoscopic Ultrasound (EUS) - Guided Celiac Plexus Neurolysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Anand Sahai MD, MSc (Epid), FRCPC, CHUM, Universite de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ND05.083
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Inoperable, Painful Pancreatic Cancer
Keywords: Pancreatic cancer; Therapy; Neurolysis
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurolysis (Active Comparator): Patients will undergo EUS followed by EUS-guided, bilateral neurolysis with bupivicaine and absolute alcohol.
  Interventions: Procedure: EUS-guided celiac plexus neurolysis
- Conventional therapy (No Intervention): EUS will be performed with no celiac plexus neurolysis.

INTERVENTIONS:
Procedure: EUS-guided celiac plexus neurolysis — Injection of 20cc of absolute alcohol + 10c of 0.5% bupivicaine on either side of the celiac axis.
  Arms: Neurolysis

SUMMARY:
Pancreatic cancer presents with pain in the majority of cases. Destruction of the celiac ganglia by ultrasound guided injection of sclerosing agents such as alcohol is sometimes used for pain that no longer responds to treatment with narcotics. The investigators compare standard narcotic treatment to celiac plexus alcohol injection (celiac plexus neurolysis) and do so in patients with early, mild pain to see if celiac plexus neurolysis is more effective than narcotics and prevents escalating narcotic use.

DETAILED DESCRIPTION:
This is a randomized, double blind, sham-controlled trial designed to evaluate the efficacy of early EUS-guided celiac plexus neurolysis (EUS-CPN). "Early" refers to the fact that, in contrast to previous CPN trials, we targeted patients with inoperable, painful pancreatic cancer in whom pain was mild and who were taking little or no narcotics. Our a priori hypotheses were that, compared to conventional management with narcotics alone, early neurolysis: 1) will better control pain related to inoperable pancreatic cancer, 2) will prevent the escalating use of narcotics associated with disease progression, 3) will improve quality of life, and 4) will improve survival. The aim our study is to test these 4 hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* previous imaging and/or the EUS examination demonstrated inoperable pancreatic cancer defined as involvement of the superior mesenteric vein, portal vein or confluence, superior mesenteric artery, celiac axis, hepatic artery, or non-regional lymphadenopathy
* a new diagnosis of pancreatic adenocarcinoma was confirmed by an on-site cytopathologist following EUS fine needle aspiration (EUS-FNA)

Exclusion Criteria:

* allergy to bupivicaine
* possible future surgical management of the tumor
* expected survival less than 3months (suspected or proven carcinomatosis or liver metastases)
* inability or unwillingness to provide informed consent prior to the EUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Absolute and relative changes in 7-point Likert-score for abdominal pain at 1 and 3 months post-randomization. Secondary endpoints were change in morphine equivalent consumption (MEQ), quality of life (DDQ-15), and overall survival. | 1 month, 3 months

SECONDARY OUTCOMES:
2. Quality of life 3. Survival | 1 month, 3 months and until death

CONTACTS AND LOCATIONS:
Overall Officials: Anand Sahai, MD, Study Director — CHUM, Universite de Montreal
Locations (1):
- CHUM, Montreal, Quebec, Canada